CLINICAL TRIAL: NCT03465267
Title: Comparing of Effects of Upper Extremity Rehabilitation on Upper Extremity Rehabilitation Robot Therapy Using Armeo Power and Armeo Spring - Randomized Controlled Trial
Brief Title: Comparisons of Two Types of Armeo Robot for Upper Extremities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2017-01-007
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Stroke
Keywords: stroke; upper extremity rehabilitation robot; stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor does not know the allocation of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Armeo power (Experimental): Armeo power robot for upper extremity
  Interventions: Device: Armeo power
- Armeo spring (Experimental): Armeo spring robot for upper extremity
  Interventions: Device: Armeo spring

INTERVENTIONS:
Device: Armeo power — Intervention with Armeo power rehabilitation robot for upper extremity (made by Hocoma), which provide assistive force.
  The intervention was done 4 weeks, 5 times/week, 30 minutes/day.
  Arms: Armeo power
Device: Armeo spring — Intervention with Armeo spring rehabilitation robot for upper extremity (made by Hocoma), which is operated only by participants, without any assistive force from robot.
  The intervention was done 4 weeks, 5 times/week, 30 minutes/day.
  Arms: Armeo spring

SUMMARY:
Comparison of two types of robot (Armeo power vs Armeo spring) for upper extremity rehabilitation on upper extremity function

DETAILED DESCRIPTION:
The purpose of this study is to compare two types of robot. The robot used in this experiment was Armeo power and Armeo spring. Armeo power could provide assistive force via motor, on the other hand, Armeo spring could not provide any assist.

Thus the results from this study might suggest usefulness of motorized robot.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Onset ≥ 3 months
* 26 ≤ Fugl-Meyer Assessment score ≤ 50
* 3 ≤ Shoulder or elbow MRC scale ≤ 4
* Shoulder or elbow flexor spasticity modified ashworth scale ≤ 1+
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* History of surgery of affected upper limb
* Fracture of affected upper limb

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Wolf motor function test | change from baseline at 4 weeks
  Change of Wolf motor function test

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Fugl-Meyer Assessment
Stroke impact scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Stroke impact scale (Health-related quality of life measurements in stroke patients)
Motor activity log | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Motor activity log
Mean velocity of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Curvature of the magnetic sensor trajectory (Kinematics of upper extremity)during reaching task
Curvature of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Curvature of the magnetic sensor trajectory (Kinematics of upper extremity during) reaching task
Jerk of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Jerk of the magnetic sensor trajectory (Kinematics of upper extremity during) reaching task
% maximal voluntary contraction of upper extremity muscles during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  surface EMG of upper extremity during reaching task
Behavioral activation system/behavioral inhibition system scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Behavioral activation system subscale, behavioral inhibition system subscale
Beck depression index | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Beck depression index
Intrinsic motivation inventory | baseline, 4 weeks after baseline, 8 weeks after baseline
  Intrinsic motivation inventory
Stroke rehabilitation motivation scale | baseline, 4 weeks after baseline, 8 weeks after baseline
  Stroke rehabilitation motivation scale

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JH, Park G, Kim HY, Lee JY, Ham Y, Hwang D, Kwon S, Shin JH. A comparison of the effects and usability of two exoskeletal robots with and without robotic actuation for upper extremity rehabilitation among patients with stroke: a single-blinded randomised controlled pilot study. J Neuroeng Rehabil. 2020 Oct 19;17(1):137. doi: 10.1186/s12984-020-00763-6. PMID 33076952